CLINICAL TRIAL: NCT00097695
Title: Randomized, Double Blind, Placebo-Controlled, Multicenter Study of a Subcutaneous Formulation of Icatibant for the Treatment of Hereditary Angioedema
Brief Title: Subcutaneous Treatment With Icatibant for Acute Attacks of Hereditary Angioedema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: JE049 #2103; FAST1 (Other: Shire HGT)
Record Dates: First submitted 2004-11-26; First posted 2004-11-29 (Estimated); Results first posted 2013-12-24 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Angioedema
Keywords: Hereditary Angioedema; C1 inhibitor deficiency; HAE; Icatibant; Bradykinin antagonist; acute attack; subcutaneous
MeSH Terms: conditions — Angioedema; Angioedemas, Hereditary | interventions — icatibant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Icatibant- Randomized (Experimental): Patients who were randomized to icatibant in the controlled phase after they had an eligible first in-study attack.
  Interventions: Drug: Icatibant
- Placebo-Randomized (Placebo Comparator): Patients who were randomized to placebo in the controlled phase after they had an eligible first in-study attack.
  Interventions: Drug: Placebo
- Controlled Open-label / laryngeal attack (Experimental): Patients with laryngeal symptoms at the baseline were not randomised but treated with icatibant open label during the controlled phase.
  Interventions: Drug: Icatibant
- Untreated Patients at the baseline (Experimental): Patients who were screened and found eligible but did not experience an angioedema attack, or had an attack that was not severe enough to merit treatment while the controlled phase was ongoing (they were not treated during the Controlled phase but treated with icatibant during the Open Label Extension Phase (OLE) )
  Interventions: Drug: Icatibant

INTERVENTIONS:
Drug: Icatibant — 30 mg (3mL) subcutaneous icatibant injection in the abdominal region
  Other Names: Brand name, Firazyr®
  Arms: Controlled Open-label / laryngeal attack; Icatibant- Randomized; Untreated Patients at the baseline
Drug: Placebo — Solution for injection, matched to study drug Single dose: 3 mL
  Arms: Placebo-Randomized

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Icatibant, a bradykinin antagonist in the treatment of acute cutaneous and/or abdominal attacks in patients with hereditary angioedema (HAE).

DETAILED DESCRIPTION:
This Phase II/III study consisted of two parts: A controlled phase and An Open label extension(OLE) phase. The controlled phase describes the double blind part of the study and was intended to evaluate the efficacy of icatibant in decreasing the time to onset of symptom relief compared with placebo for the first treated cutaneous and/or abdominal attack in randomised patients. Patients experienced a laryngeal attack were not randomised, but treated with open label icatibant according to the controlled phase procedures and assessments. The outcome of this group was to be reported descriptively. After treatment of the first attack in the controlled phase, the patients were eligible to enter the OLE phase. In the OLE phase, patients who experienced angioedema attacks severe enough to warrant treatment were to be treated with s.c. icatibant as appropriate until the end of the study.The OLE phase became a modified open label extension where all 56 patients who had been randomised and the last randomised patient had concluded the double-blind phase. The modified open label extension period permitted treatment for patients who were screened and found eligible but did not experience an angioedema attack, or had an attack that was not severe enough to merit treatment while the double blind phase was still ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years;
* Documented diagnosis of HAE Type I or II (confirmed complement 1 esterase inhibitor [C1-INH] deficiency);
* Current edema be in the cutaneous, abdominal and/or laryngeal areas;
* Current edema be moderate to severe according to the investigator's Symptom Score.

Exclusion Criteria:

* Diagnosis of angioedema other than HAE, for example, acquired angioedema (AAE);
* Participation in a clinical trial of another investigational medicinal product (IMP) within the past month;
* Treatment with any pain medication since onset of the current edema attack;
* Treatment with replacement therapy, including C1-INH products (e.g. human C1-INH preparations), less than 3 days from onset of the current edema attack;
* Treatment with ACE inhibitors (e.g. Lotensin, Prinivil, Accupril);
* Evidence of severe, symptomatic coronary artery disease based on medical history or screening examination;
* Serious concomitant illnesses that the physician considers to be a contraindication for participation in the trial;
* Pregnancy and/or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2004-12-28 (Actual); Primary Completion 2006-07-17 (Actual); Study Completion 2006-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Georgetown University Hospital, Lombardi Cancer Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Malbran A, Riedl M, Ritchie B, Smith WB, Yang W, Banerji A, Hebert J, Gleich GJ, Hurewitz D, Jacobson KW, Bernstein JA, Khan DA, Kirkpatrick CH, Resnick D, Li H, Fernandez Romero DS, Lumry W. Repeat treatment of acute hereditary angioedema attacks with open-label icatibant in the FAST-1 trial. Clin Exp Immunol. 2014 Aug;177(2):544-53. doi: 10.1111/cei.12358. PMID 24749847
- [Derived] Cicardi M, Banerji A, Bracho F, Malbran A, Rosenkranz B, Riedl M, Bork K, Lumry W, Aberer W, Bier H, Bas M, Greve J, Hoffmann TK, Farkas H, Reshef A, Ritchie B, Yang W, Grabbe J, Kivity S, Kreuz W, Levy RJ, Luger T, Obtulowicz K, Schmid-Grendelmeier P, Bull C, Sitkauskiene B, Smith WB, Toubi E, Werner S, Anne S, Bjorkander J, Bouillet L, Cillari E, Hurewitz D, Jacobson KW, Katelaris CH, Maurer M, Merk H, Bernstein JA, Feighery C, Floccard B, Gleich G, Hebert J, Kaatz M, Keith P, Kirkpatrick CH, Langton D, Martin L, Pichler C, Resnick D, Wombolt D, Fernandez Romero DS, Zanichelli A, Arcoleo F, Knolle J, Kravec I, Dong L, Zimmermann J, Rosen K, Fan WT. Icatibant, a new bradykinin-receptor antagonist, in hereditary angioedema. N Engl J Med. 2010 Aug 5;363(6):532-41. doi: 10.1056/NEJMoa0906393. PMID 20818888

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients must have an eligible HAE attack to be randomized.64 patients were in the controlled phase(27icatibant,29 placebo,8subjects with laryngeal attacks were treated with open label icatibant).A total of 72 were treated in the open label phase(20 entered directly into the OLE phase+ 52 from the controlled phase).
Groups:
- Randomized -Icatibant: Patients who were randomized to icatibant in the controlled phase after they had an eligible first in-study attack.
- Randomized -Placebo: Patients who were randomized to placebo in the controlled phase after they had an eligible first in-study attack.
- Untreated Patients at the Baseline: Patients who were screened and found eligible but did not experience an angioedema attack, or had an attack that was not severe enough to merit treatment while the controlled phase was ongoing.
Period: The Controlled Phase
Arm/Group | Randomized -Icatibant | Randomized -Placebo | Controlled Open-label / Laryngeal Attack | Untreated Patients at the Baseline
Started | 27 | 29 | 8 | 20
Completed | 23 | 26 | 3 | 0 (Patients screened and found eligible but did not have HAE attack or attack was not severe enough)
Not Completed | 4 | 3 | 5 | 20
Period: The Open Label Extension (OLE) Phase
Arm/Group | Randomized -Icatibant | Randomized -Placebo | Controlled Open-label / Laryngeal Attack | Untreated Patients at the Baseline
Started | 23 | 26 | 3 | 20
Completed | 10 | 11 | 1 | 15
Not Completed | 13 | 15 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Controlled Open-label / Laryngeal Attack: patients who received first treatment Open-Label due to laryngeal symptoms
- Total: Total of all reporting groups
Arm/Group | Randomized -Icatibant | Randomized -Placebo | Controlled Open-label / Laryngeal Attack | Untreated Patients at the Baseline | Total
Number analyzed (Participants) | 27 | 29 | 8 | 20 | 84
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.8 (9.81) | 34.9 (11.37) | 47.1 (13.86) | 37.4 (11.48) | 36.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 5 | 15 | 57
  Male | 11 | 8 | 3 | 5 | 27

OUTCOME MEASURES:

1. Primary Outcome: Time to Onset of Symptom Relief (TOSR)
Description: The primary efficacy endpoint was TOSR assessed by the patient using a Visual Analogue Scale (VAS). The VAS is a scale used to measure intensity of each symptom of the attack at baseline and at the pre-determined time points throughout treatment period. It consists of a horizontal 10cm line, with the 0 point corresponding to a state where patient experiences no symptoms at all and the 10cm point represents the worst symptoms ever experienced by patient. The patient indicates his/her current state of symptoms by drawing a mark across the horizontal line. TOSR was defined as the time between time of injection to time of first documented onset of symptom relief for the 3 primary symptoms: cutaneous swelling, cutaneous skin, and abdominal pain. The primary symptom was based on the type of attack. For abdominal attacks, the single primary symptom was abdominal pain. For cutaneous attacks, the single primary symptom was either skin swelling or skin pain, whichever was most severe.
Time Frame: 5 days
Population: Time to onset of symptom relief - Controlled phase - ITT population (patients experiencing moderate to very severe acute cutaneous and/or abdominal HAE attacks)
Measure: Median (Inter-Quartile Range); unit: Hours
Groups:
- Randomized -Icatibant: 27 Patients were randomized to icatibant in the controlled phase after they had an eligible first in-study attack.
- Randomized -Placebo: 29 Patients were randomized to placebo in the controlled phase after they had an eligible first in-study attack.
Arm/Group | Randomized -Icatibant | Randomized -Placebo
Number analyzed (Participants) | 27 | 29
Hours | 2.5 [1.1 to 6.0] | 4.6 [1.8 to 10.2]
Statistical Analysis 1: Comparison: Randomized -Icatibant vs Randomized -Placebo; Test type: Superiority or Other; p = 0.142, Wilcoxon version of the log-rank test; The Wilcoxon version of the log-rank test of SAS was used to calculate statistical significance between p- vs icatibant group and placebo group

2. Secondary Outcome: Time to Regression (Start of Improvement) According to Patient
Description: This parameter assessed the time to regression (start of improvement) of observable(visible) symptoms according to the patients. Patients were asked "Report date and time when you feel that your symptoms start to improve".
Time Frame: 5 days
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Randomized -Icatibant | Randomized -Placebo
Number analyzed (Participants) | 27 | 29
Hours | 0.8 [0.5 to 2.0] | 16.9 [3.2 to NA] — 14 patients were censored in the placebo group; these patients were censored as no data for time to regression (start of improvement) according to the patient were documented within the observation period.
Statistical Analysis 1: Comparison: Randomized -Icatibant vs Randomized -Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon version of the log-rank test; The median time to onset is calculated using Kaplan-Meier methodology. The Wilcoxon version of the log-rank test of SAS is used

3. Secondary Outcome: Time to Almost Complete Symptom Relief
Description: The time to almost complete symptom relief was defined as a score between 0 and 10 mm on the VAS for at least 3 consecutive measurements for all symptom.
Time Frame: 5 days
Measure: Median (Inter-Quartile Range); unit: Hours
Groups:
- Randomized Control Trial-icatibant: 27 Patients were randomized to icatibant in the controlled phase after they had an eligible first in-study attack.
- Randomized Control Trial-placebo: 29 Patients were randomized to placebo in the controlled phase after they had an eligible first in-study attack.
Arm/Group | Randomized Control Trial-icatibant | Randomized Control Trial-placebo
Number analyzed (Participants) | 27 | 29
Hours | 8.5 [2.5 to 31.5] | 19.4 [10.2 to 55.7]
Statistical Analysis 1: Comparison: Randomized Control Trial-icatibant vs Randomized Control Trial-placebo; Test type: Superiority or Other; p = 0.079, Wilcoxon version of the log-rank test; The median time to almost complete symptom relief was calculated using Kaplan-Meier methodology.The Wilcoxon version of the log-rank test of SAS used

ADVERSE EVENTS:
Time Frame: An AE was assigned to the controlled phase if the event start date was between the first treatment of the first attack and the first treatment in the OLE phase.
Groups:
- Controlled Phase- Icatibant (Randomized Subjects ): Patients who were randomized to icatibant in the controlled and experienced adverse events while participating in the controlled phase.
- Controlled Phase- Placebo (Randomized Subjects: Patients who were randomized to placebo in the controlled phase and experienced adverse events while participating in the controlled phase.
- Controlled Phase- Icatibant (Subjects w/ Laryngeal Attack): This represents adverse events during the controlled phase that were experienced by Patients with laryngeal symptoms at the baseline and were treated with open label icatibant during the controlled phase.
- Open Label Extension Phase- Icatibant (Previously Randomized): Patients who were randomized to either icatibant or placebo in the controlled phase and experienced adverse events while participating in the open label extension phase.
- Open Label Extension -Icatibant (Subjects w/ Laryngeal Attack): This represents adverse events during the open label extension phase that were experienced by Patients with laryngeal symptoms at the baseline and got treated with open label icatibant during the controlled phase.
- Open Label Extension Phase(Untreated Patients at the Baseline): This represents adverse events experienced by Patients who were screened and found eligible but did not experience an angioedema attack, or had an attack that was not severe enough to merit treatment while the controlled phase was ongoing.
Arm/Group | Controlled Phase- Icatibant (Randomized Subjects ) | Controlled Phase- Placebo (Randomized Subjects | Controlled Phase- Icatibant (Subjects w/ Laryngeal Attack) | Open Label Extension Phase- Icatibant (Previously Randomized) | Open Label Extension -Icatibant (Subjects w/ Laryngeal Attack) | Open Label Extension Phase(Untreated Patients at the Baseline)
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/29 | 1/8 | 3/49 | 0/3 | 0/20
Other Adverse Events (participants affected / at risk) | 12/27 | 19/29 | 6/8 | 39/49 | 3/3 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Controlled Phase- Icatibant (Randomized Subjects ) (N=27) | Controlled Phase- Placebo (Randomized Subjects (N=29) | Controlled Phase- Icatibant (Subjects w/ Laryngeal Attack) (N=8) | Open Label Extension Phase- Icatibant (Previously Randomized) (N=49) | Open Label Extension -Icatibant (Subjects w/ Laryngeal Attack) (N=3) | Open Label Extension Phase(Untreated Patients at the Baseline) (N=20)
HAE attack (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Controlled Phase- Icatibant (Randomized Subjects ) (N=27) | Controlled Phase- Placebo (Randomized Subjects (N=29) | Controlled Phase- Icatibant (Subjects w/ Laryngeal Attack) (N=8) | Open Label Extension Phase- Icatibant (Previously Randomized) (N=49) | Open Label Extension -Icatibant (Subjects w/ Laryngeal Attack) (N=3) | Open Label Extension Phase(Untreated Patients at the Baseline) (N=20)
Dizziness (Investigations) | 2 | 1 | 0 | 0 | 1 | 0
Headache/Migraine (Nervous system disorders) | 0 | 2 | 2 | 0 | 2 | 1
Hereditary angioedema (Congenital, familial and genetic disorders) | 4 | 5 | 4 | 17 | 1 | 5 — HAE attacks were over-reported as AEs as some investigators reported new attacks as AEs in addition to worsening of attacks in Icatibant treated patients.
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Infections (Infections and infestations) | 4 | 4 | 1 | 20 | 0 | 7
Administration site conditions (General disorders) | 3 | 4 | 0 | 11 | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less